CLINICAL TRIAL: NCT00429858
Title: Individualized Management of Pancreatic Cancer With Targeted Therapeutics (IMPACTT): A Phase II Clinical Trial
Brief Title: Gemcitabine and S-1 for Locally Advanced Unresectable or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study accrual rate is very slow, it was mandated by NCI to be terminated.
Sponsor: Andrew Ko (Other)
Collaborators: Eli Lilly and Company (Industry); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Ko, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06456; NCI-2011-01215 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); UCSF-H12191-29556-01 (Other: UCSF California CHR Approval #)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); titanium silicide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Targeted therapy group (Experimental): Gemcitabine monotherapy until disease progression, followed by gemcitabine + S-1
  Interventions: Drug: S-1; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: S-1 — S-1 is given as follows: 25 mg/m2 bid on days 1-7 and 15-21 of the cycle (28 days)
  Other Names: tegafur-gimeracil-oteracil potassium; TS-1; TS-ONE
Drug: gemcitabine hydrochloride — Patients will receive gemcitabine at a dose of 1,000 mg/m2 i.v. at a fixed-dose rate (FDR) infusion of 10 mg/m2/minute (100 minutes), once a week for 3 consecutive weeks, followed by one week rest. Each 4 week period is referred to as a treatment cycle
  Other Names: Gemzar

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer. It may also help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial is studying gene expression in predicting treatment response in patients receiving gemcitabine and S-1 for locally advanced unresectable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate intratumoral expression level of ribonucleotide reductase subunit 1 (RRM1) with response to gemcitabine hydrochloride therapy in patients with locally advanced unresectable or metastatic adenocarcinoma of the pancreas.

Secondary

* Correlate intratumoral expression levels of other genes (e.g., deoxycytidine kinase [dCK], equilibrative nucleoside transporter 1 [ENT1], and concentrative nucleoside transporters 1 and 3 [CNT1 and CNT3]) with response in these patients.
* Determine, preliminarily, the median survival of these patients, using a therapeutic strategy entailing sequential addition of agents and decision making based on early CA 19-9 biomarker response.
* Determine the safety of this approach.
* Determine the percentage of patients classified as potential biomarker responders.
* Determine the time to progression with each successive line of treatment.
* Determine the proportion of patients with ≥ 25% decline in CA 19-9 biomarker (i.e., biomarker response) with each successive line of treatment.

Tertiary

* Identify other genes that may mediate sensitivity to gemcitabine hydrochloride, S-1, and other agents with activity in pancreatic cancer.
* Determine the frequency of host genetic polymorphisms in various nucleoside transporters.

OUTLINE: This is a multicenter.

* Initial treatment (gemcitabine hydrochloride alone): Patients receive gemcitabine hydrochloride IV over 100 minutes on days 1, 8, and 15. CA 19-9 levels are assessed in weeks 1 and 3 of each course. Patients who are biomarker responders continue to receive treatment with gemcitabine hydrochloride alone. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are no longer biomarker responders or show other evidence of disease progression proceed to therapy comprised of gemcitabine hydrochloride and S1.
* Gemcitabine hydrochloride and S-1 treatment: Patients receive gemcitabine hydrochloride IV over 100 minutes on days 1 and 15 and oral S-1 twice daily on days 1-7 and 15-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo core needle tumor biopsy and fine-needle aspiration at baseline. Tissue samples are analyzed for correlation between transcript and protein expression by immunohistochemistry and for expression of genes and gene products that may mediate sensitivity to gemcitabine hydrochloride (RRM1, ENT1, CNT1 and 3, dCK); S-1, thymidine phosphorylase [TP], TS, DPD, and ORPT; and other anticancer treatments (ERCC-1, epidermal growth factor receptor, GSK-3β) by reverse-transcriptase polymerase chain reaction. Tissue samples are also analyzed by microarray and comparative genomic hybridization to identify new genes that may predict chemotherapeutic response or mediate sensitivity to anticancer therapy. Mutational status of KRAS and p53 gene are also assessed.

Blood samples are collected at baseline and are analyzed by genotyping assays to identify polymorphic variants of select genes.

After completion of study treatment, patients are followed monthly.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria

* Adenocarcinoma of the pancreas that is already or will be histologically or cytologically proven.
* Patients must have either locally advanced (unresectable) or metastatic disease.
* Radiographically measurable disease is not required.
* No prior therapy for advanced pancreatic cancer. Treatment given in the adjuvant setting (radiation and/or chemotherapy, given either concurrently or systemically) does not count as prior therapy as long as progressive disease occurs > 6 months following completion of treatment.
* Greater than or equal to 18 years of age.
* ECOG performance status of 0 or 1 (See Appendix D).
* Laboratory criteria:
* ANC > 1500/µL
* Platelet count > 100,000/µL
* Hemoglobin > 9 g/dL (may be transfused or receive epoetin alfa to maintain or exceed this level)
* INR < 1.5 (except those subjects who are receiving full-dose warfarin
* Total bilirubin < 2.0 mg/dL
* AST or ALT < 5 times upper limit of normal for subjects with documented liver metastases; < 2.5 times the upper limit of normal for subjects without evidence of liver metastases
* Serum creatinine < 2.0 mg/dL
* Serum CA19-9 > 2X upper limits of normal.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Women or men of reproductive potential must agree to use an effective contraceptive method during treatment and for 6 months afterwards.

Exclusion criteria

* Inability to comply with study and/or follow-up procedures
* Disease determined to be not amenable to biopsy upon review of radiographs by the oncologist and/or interventional radiologist.
* Clearly resectable disease in a patient who is an appropriate operative candidate.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Prior systemic therapy for advanced pancreatic cancer
* Pregnant (positive pregnancy test) or lactating
* Use of anti-neoplastic or anti-tumor agents not part of the study therapy, including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy, is not permitted while participating in this study.
* Use of concurrent investigational agents is not permitted.

S-1 Specific Exclusion Criteria

* Is receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:
* Sorivudine, brivudine, uracil, dipyridamole, cimetidine, and folinic acid (may enhance S-1 activity).
* Allopurinol (may diminish S-1 activity).
* Phenytoin (S-1 may enhance phenytoin activity).
* Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 and flucytosine activity).
* Pilocarpine (may inhibit cytochrome P-450 enzyme 2A6 activity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2010-01-20 (Actual); Study Completion 2010-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Targeted Therapy Group
Started | 21
Completed | 19
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Study Termination | 1

BASELINE CHARACTERISTICS:
Population: Patient demographic data was retained electronically when transferred from legacy system.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 2
  50-59 years old | 5
  60-69 years old | 11
  70-79 years old | 2
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Correlate Intratumoral Expression Level of Ribonucleotide Reductase Subunit 1 (RRM1) With Response to Gemcitabine in Patients With Advanced Pancreatic Cancer.
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between RRM1 and response to gemcitabine. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of RRM1 and response to gemcitabine, a value of 0 indicating no association between RRM1 and response to gemcitabine, and a value of +1 indicating a positive linear association of RRM1 and response to gemcitabine.
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlate Intratumoral Expression Levels of Other Genes, Including Deoxycytidine Kinase (dCK), Equilibrative Nucleoside Transporter 1 (ENT1) and Concentrative Nucleoside Transporters 1 and 3 (CNT1 and CNT3), With Response to Gemcitabine.
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between deoxycytidine kinase (dCK), equilibrative nucleoside transporter 1 (ENT1) and concentrative nucleoside transporters 1 and 3 (CNT1 and CNT3), with response to gemcitabine in a table format. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of intratumoral expression levels and response to gemcitabine, a value of 0 indicating no association between intratumoral expression levels and response to gemcitabine, and a value of +1 indicating a positive linear association of intratumoral expression levels and response to gemcitabine.
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlate Intratumoral Expression Levels of Thymidylate Synthase (TS), Thymidine Phosphorylase (TP), Dihydropyrimidine Dehydrogenase (DPD), Orotate Phosphoribosyltransferase (ORPT) With Response to the Combination of Gemcitabine/S-1.
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between intratumoral expression levels of thymidylate synthase (TS), thymidine phosphorylase (TP), dihydropyrimidine dehydrogenase (DPD), orotate phosphoribosyltransferase (ORPT) with response to the combination of gemcitabine/S-1 in a table format. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of intratumoral expression levels and the combination of gemcitabine/S-1, a value of 0 indicating no association between intratumoral expression levels and response to the combination of gemcitabine/S-1, and a value of +1 indicating a positive linear association of intratumoral expression levels and response to the combination of gemcitabine/S-1.
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Median Overall Survival
Description: Overall survival will be defined from the date of receiving the first treatment until death
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients With Dose Modifications
Description: Treatment-related toxicities resulting in a dose modification be classified using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 will be tabulated.
Time Frame: 8 weeks after 6th patient is enrolled
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Patients Classified as Potential Biomarker Responders
Description: Defined as the percentage of patients who will be categorized as potential biomarker responders if their CA19-9 has declined by > 10 % from peak value (peak value may have been at either week 1 or 3) during the initial gemcitabine monotherapy phase
Time Frame: Assessed after the first 5 weeks of treatment
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Time to Progression
Description: Time to progression will be summarized according to the method of Kaplan and Meier
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Patients With at Biomarker Response
Description: A biomarker response for any given line of therapy is defined as patients with a baseline CA19-9 level > 75 units per cubic centimeter (U/cc) who demonstrate a > 25% decline in their peak CA19-9 level, sustainable for at least 2 consecutive measurements
Time Frame: Up to 2 years
Population: Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Data for non-serious adverse events was not migrated from legacy clinical trials management system, due to the study closure with the University of California, San Francisco (UCSF) institutional review board (IRB) prior to system migration. Historical records were discarded in accordance with university record retention policy.
Arm/Group | Targeted Therapy Group
All-Cause Mortality (participants affected / at risk) | 7/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Therapy Group (N=21)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomitting (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Pain, NOS (General disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemorrhage, GI - Duodenum (Gastrointestinal disorders) | 1 (1)
Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Historical records were discarded in accordance with university record retention policy. Data electronically archived to the current clinical trial management system has been reported where possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes